CLINICAL TRIAL: NCT05329142
Title: ASSIST: A Surveillance Study of Illicit Substance Toxicity - Clinical Characterisation and Toxicological Analysis of Emergency Department Presentations in Glasgow
Brief Title: ASSIST: A Surveillance Study of Illicit Substance Toxicity
Acronym: ASSIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: Public Health Scotland (Unknown)
Responsible Party: Sponsor
Other Study IDs: GN21AE239
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Overdose, Drug; Drug Use; Drug Abuse; Drug Toxicity; Drug Effect; Illicit Drug Use; Illicit Drug Overdose; Illicit Drug Intoxication
MeSH Terms: conditions — Drug Overdose; Substance-Related Disorders; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A surplus sample of blood taken as part of usual care biochemistry sample from selected patients will be analysed by way of Mass Spectrometry.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 1: Usual Care clinical data:: The patient will firstly be identified as having attended the ED due to acute illicit drug toxicity and must fit the inclusion and exclusion criteria. The research team will complete the electronic Case Report Form (eCRF), which will include defined data.
- Stage 2: Surplus sampling Mass Spectrometry: The research team will select patients with acute moderate / severe toxicity, which will be defined as those requiring at least one of:
  * Patient admitted to hospital due to acute illicit drug toxicity
  * Pre-hospital cardio/pulmonary resuscitation
  * Any part of patient's ED care was in the Resuscitation area of the ED
  * Patient died in the ED or within 72 hours
  A surplus sample of the standard of care SST sample from this group will be analysed by way of Mass Spectrometry.
  Interventions: Diagnostic Test: Surplus sample toxicology analysis

INTERVENTIONS:
Diagnostic Test: Surplus sample toxicology analysis — Anonymised surplus blood sample will be analysed for drugs and their metabolites by way of Mass Spectrometry and LGC Group, Cambridge.
  Groups: Stage 2: Surplus sampling Mass Spectrometry

SUMMARY:
There is a drug-related death crisis in Scotland. This study aims to collaborate with Public Health Scotland in order to assess the feasibility of introducing a surveillance system to the Emergency Department to highlight illicit drug-related attendances. This will utilise both clinical data and toxiclogical analysis of anonymised samples. The data will inform of prevalence, trend data and utcome of ED patients attending with acute illict drug toxicity.

DETAILED DESCRIPTION:
The purpose of this research is to establish the introduction of a robust toxicology surveillance system in the Emergency Department (ED) in order to inform public health interests. The study will explore the feasibility of reporting characteristics and causative agents of patients attending hospital as an emergency due illicit substance use. The term illicit substance used during this study encompasses any substance which is not prescribed to the individual and is a controlled drug as per the Misuse of Drugs act 1971 and Misuse of Drugs Regulations 2001.

The study will look at standard care clinical data from all individuals attending the Emergency Department due to acute illicit drug toxicity. Surplus blood samples will be anonymised and analysed for toxicological profiling.

The study will allow identification of emerging drug trends and will be shared contemporaneously with Public Health Scotland and inform the Scottish Government of current incidences to inform public health measures to tackle the drugs death crisis.

ELIGIBILITY:
Inclusion Criteria:

* Age >16
* Patient attending QEUH ED directly relating to acute illicit drug use
* Patients with reported acute illicit drug use toxicity who are unwell before they are seen in the Emergency Department but appear well in the ED should also be included

Exclusion Criteria:

* Condition more likely due to cause other than acute illicit drug use
* Condition due to withdrawal of drugs / alcohol
* Condition primarily related to alcohol use and no evidence of acute illicit drug use
* Attendance is due to complication of previous drug use - i.e., BBV / infected injection site (without acute drug toxicity)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stage 1: All adult patients attending Queen Elizabeth University Hospital ED due to acute illicit substance use. The target is 1000 patients.
  Stage 2: Patients from stage 1 with moderate / severe toxicity as described in section 7.1. The target number of participants in this study is 500.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2023-08-19 (Estimated); Study Completion 2023-08-19 (Estimated)

PRIMARY OUTCOMES:
Proportion of full data sets and toxicology analysis for all patient attending the ED due to acute illicit drug toxicity | 1 year
  Objective:
  Assess the feasibility of prospective surveillance of Emergency Department presentations relating to acute illicit drug toxicity
  Outcome measure:
  Proportion of full data sets and toxicology analysis for all patient attending the ED due to acute illicit drug toxicity

SECONDARY OUTCOMES:
Clinical phenotyping of patients attending due to acute illicit drug toxicity compared to reported / presumed drug taken | 1 year
  Objective:
  Describe the clinical characteristics and reported / presumed toxicological profile of drug related presentations to the Emergency Department
  Outcome measure:
  Clinical phenotyping of patients attending due to acute illicit drug toxicity compared to reported / presumed drug taken
Proportion of patients who fit stage 2 criteria with biological sample mass spectrometry toxicology analysis | 1 year
  Objective:
  Establish the feasibility of ED presentation toxicological surveillance by anonymised surplus sample mass spect analysis
  Outcome Measure:
  Proportion of patients who fit stage 2 criteria with biological sample mass spectrometry toxicology analysis
Production of frequency and trend data to deliver to Public Health Scotland | 1 year
  Objective:
  Describe the frequency and trends of drug related presentations to the ED, both clinically and by biological sample analysis
  Outcome measure:
  Production of frequency and trend data to deliver to Public Health Scotland
Proportion of illicit drug reported to have been taken and proportion of clinician presumed drug taken accurately matching toxicology analysis | 1 year
  Objective:
  Assess the accuracy of reported / clinician presumptive toxidrome diagnosis compared to biological sample analysis
  Outcome Measure:
  Proportion of illicit drug reported to have been taken and proportion of clinician presumed drug taken accurately matching toxicology analysis
Production of automated pre-defined data capture, recording and auditing for the routine processing of drug related ED presentations that includes toxicological information | 1 year
  Objective:
  Develop a framework to standardise data capture, recording and auditing for the routine processing of drug related ED presentations that includes toxicological information
  Outcome measure:
  Production of automated pre-defined data capture, recording and auditing for the routine processing of drug related ED presentations that includes toxicological information
Share learning and data with Scottish Government, PHS and other NHS boards to inform national scale up | 1 year
  Objective:
  Identify and compare options for national scale up - including the use of existing hospital toxicology facilities and additional services
  Outcome measure:
  Share learning and data with Scottish Government, PHS and other NHS boards to inform national scale up

CONTACTS AND LOCATIONS:
Overall Officials: David J Lowe, MBChB BMSc FRCEM, Principal Investigator — NHS GGC R&I Non Commerical (Sponsor) Research Coordinator
Locations (1):
- Queen Elizabeth University Hospital, NHS GGC, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] UK Public General Acts. Misuse of Drugs Act 1972 Schedule 2. Available from legislation.gov.uk. Accessed 25/02/2022
- [Background] The Misuse if Drugs Regulations 2001, Dangerous Drugs. Available from legislation.giv.uk. Accessed 25/02/2022.
- [Background] EMCDDA. European Drug Report, trends and Developments 2021. Available from https://www.emcdda.europa.eu/system/files/publications/13838/TDAT21001ENN.pdf accessed 14/02/2022
- [Background] National Records of Scotland. Drug-related deaths in Scotland in 2020, published 30/07/21. Available from https://www.nrscotland.gov.uk. Accessed 14/02/2022.
- [Background] Public Health Scotland, Drug-related Hospital Statistics, Scotland 2019 - 2020. Published 15/06/2021. Available from https://publichealthscotland.scot/. Accessed 14/02/2022
- [Background] Scottish Government. Evidence-Based Strategies for Preventing Drug-Related Deaths in Scotland, Our Emergency Response. January 2020. Available from https://www.gov.scot/. Accessed 10/02/2021
- [Background] Di Rico R, Nambiar D, Stoove M, Dietze P. Drug overdose in the ED: a record linkage study examining emergency department ICD-10 coding practices in a cohort of people who inject drugs. BMC Health Serv Res. 2018 Dec 5;18(1):945. doi: 10.1186/s12913-018-3756-8. PMID 30518362
- [Background] EMCDDA. Drug-related deaths and mortality in Europe. Update from EMCDDA expert network July 2019. Available from https://www.emcdda.europa.eu. Accessed 09/02/2020
- [Background] European Monitoring Centre for Drugs and Drug Addiction. (2016) Health responses to new psychoactive substances. Available from http://www.emcdda.europa.eu/system/files/publications/2812/TD0216555ENN.pdf. Accessed 15/02/2022
- [Background] European Monitoring Centre for Drugs and Drug Addiction (2021), European Drug Report 2021: Trends and Developments, Publications Office of the European Union, Luxembourg.
- [Background] Office for National Statistics. Drug misuse in England and Wales: year ending March 2020 09/12/2020. Accessed 16/02/2022
- [Background] Deaths mentioning a new psychoactive substance by broad age-group, England and Wales, 2011 to 2015 registrations. 18 January 2017. Available from: https://www.ons.gov.uk/peoplepopulationandcommunity/birthsdeathsandmarriages/deaths/adhocs/06556deathsmentioninganewpsychoactivesubstancebybroadagegroupenglandandwales2011to2015registrations. Accessed 19/12/2018
- [Background] Adams AJ, Banister SD, Irizarry L, Trecki J, Schwartz M, Gerona R. "Zombie" Outbreak Caused by the Synthetic Cannabinoid AMB-FUBINACA in New York. N Engl J Med. 2017 Jan 19;376(3):235-242. doi: 10.1056/NEJMoa1610300. Epub 2016 Dec 14. PMID 27973993
- [Background] Seywright A, Torrance HJ, Wylie FM, McKeown DA, Lowe DJ, Stevenson R. Analysis and clinical findings of cases positive for the novel synthetic cannabinoid receptor agonist MDMB-CHMICA. Clin Toxicol (Phila). 2016 Sep;54(8):632-7. doi: 10.1080/15563650.2016.1186805. Epub 2016 May 23. PMID 27213960
- [Background] Hikin L, Smith PR, Ringland E, Hudson S, Morley SR. Multiple fatalities in the North of England associated with synthetic fentanyl analogue exposure: Detection and quantitation a case series from early 2017. Forensic Sci Int. 2018 Jan;282:179-183. doi: 10.1016/j.forsciint.2017.11.036. Epub 2017 Nov 29. PMID 29216524
- [Derived] Dunlop LC, Craik V, Jarvie N, Hudson S, Walters M, Dear JW, Lowe DJ. Clinical characterisation of the novel benzodiazepine bromazolam-data from the ASSIST (A Surveillance Study of Illicit Substance Toxicity) study. Clin Toxicol (Phila). 2025 Nov;63(11):838-848. doi: 10.1080/15563650.2025.2524078. Epub 2025 Jul 28. PMID 40719187